CLINICAL TRIAL: NCT00979849
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled AZD8683 After Single Ascending Doses in Healthy Male Subjects
Brief Title: AZD8683 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, MSD
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1883C00001
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
Keywords: safety; tolerability; healthy; inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- A (Experimental): AZD8683
  Interventions: Drug: AZD8683
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8683 — Solution for nebulisation, inhaled. Each subject will receive a single-dose of AZD8683 or placebo. Starting dose 1 ug (lung deposited dose) with up to 8 dose escalation not exceeding AstraZeneca pre-defined exposure limits.
  Arms: A
Drug: Placebo — Solution for nebulisation, inhaled
  Arms: B

SUMMARY:
The aim of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD8683 following single ascending dose administrations in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examinations
* Use any prescribed or non-prescribed medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | Frequent sampling occasions during study days, before and up to 48 h after dosing, and at a follow-up visit 7-13 days after dosing.

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration (Cmax), time to Cmax (tmax), terminal rate constant (λz), terminal half-life (t½λz) | Frequent sampling occasions during study days, before and up to 48 h after dosing.
Pharmacokinetics: Area under the plasma concentration-time curve from zero to the time of the last measurable concentration (AUC(0-t)) and from zero to infinity (AUC), apparent plasma clearance (CL/F) | Frequent sampling occasions during study days, before and up to 48 h after dosing.
Pharmacokinetics: Apparent volume of distribution during terminal phase (Vz/F), mean residence time (MRT), amount of drug excreted unchanged (Ae; % dose), and renal clearance (CLR). | Frequent sampling occasions during study days, before and up to 48 h after dosing.
Pharmacodynamics: Lung function by spirometry (forced expiratory volume in the first second [FEV1] and forced vital capacity [FVC]), blood pressure, pulse, QTc, and heart rate. | Frequent sampling occasions during study days, before and up to 48 h after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Gurdrun Schwabe, Study Director — AstraZeneca R&D Lund; Sylvan Hurewitz, Principal Investigator — AstraZeneca CPU, Philadelphia
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States